CLINICAL TRIAL: NCT04787237
Title: Immediate Implant Placement Using Vestibular Socket Therapy Versus Early Implant Placement Using Buser's Technique for Managing Type 2 Extraction Sockets: A Randomized Clinical Trial
Brief Title: Vetsibular Socket Therapy Versus Buser's Technique
Acronym: VST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Iman Abd-ElWahab Radi, PhD, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0010558
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Dental Implant Failed

STUDY DESIGN:
Intervention Model Description: randomized clinical trial, blinded
Who Masked: Outcomes Assessor
Masking Description: AE and IR were responsible for measuring the outcomes and they were blinded to the treatments, since they were not involved in the treatment The statistician was also blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibulart socket therapy and immediate implants (Experimental): A subperiosteal tunnel was created connecting the socket orifice and the vestibular access incision using periotomes and micro periosteal elevators (. Implant fixture were then inserted . A flexible cortical membrane shield that is made of cortical bone of heterologous origin was introduced from the vestibular access incision reaching 1 mm below the socket orifice through the tunnel then stabilized using a membrane tack or a micro screw to the alveolar bone apical to the base of the socket . The socket gap between the implant and the shield was then packed thoroughly with particulate bone graft
  Interventions: Other: VST and immediate implants
- Buser's technique and early implant placement (Active Comparator): In Buser's group early implant placement, the failing tooth was extracted atraumatically using a periotome. A collagen plug was placed to stabilize the wound clot. A healing period of 4-8 weeks was followed. Then an open flap implant surgery using a triangular flap design was cut. Implant was then placed under the crest of the palatal bone. A healing abutment was then attached. Contour augmentation was done using autogenous bone chips mixed with saline and bone conditioned medium (BCM) added to bioss bone granules to activate it.
  Interventions: Other: Buser technique and early implants placement

INTERVENTIONS:
Other: VST and immediate implants — One-cm long vestibular access incision was made using a 15c blade 3-4 mm apical to the mucogingival junction at the related socket . A subperiosteal tunnel was created connecting the socket orifice and the vestibular access incision using periotomes and micro periosteal elevators (. Implant fixture were then inserted after drilling to its pre-planned location 3-4 mm apical to socket base with adequate primary stability achieved using a torque wrench reaching 30 Ncm torque . A flexible cortical membrane shield that is made of cortical bone of heterologous origin of 0.6 mm thickness was hydrated and then trimmed and introduced from the vestibular access incision reaching 1 mm below the socket orifice through the tunnel . The socket gap between the implant and the shield was then packed thoroughly with particulate bone graft
  Other Names: VST
  Arms: Vestibulart socket therapy and immediate implants
Other: Buser technique and early implants placement — In Buser's group early implant placement, the failing tooth was extracted atraumatically using a periotome. A collagen plug was placed to stabilize the wound clot. A healing period of 4-8 weeks (depending on the size of the extracted tooth) was followed. Then an open flap implant surgery using a triangular flap design was cut. After preparing the implant bed, the site was irrigated using normal saline. A healing abutment was then attached. Contour augmentation was done using autogenous bone chips mixed with saline and bone. A non-cross liked membrane was then placed, after being soaked with BCM. Finally, the healing abutment was removed and the flap was released to allow for its suturing.
  Other Names: contour augmentation and early implant placement
  Arms: Buser's technique and early implant placement

SUMMARY:
immediate implant placement using the VST was compared to early implant placement protocol using Buser's technique regarding implant survival, changes in labial plate thickness and soft tissue height after 1 year of implant placement

DETAILED DESCRIPTION:
Preoperative procedures A preoperative radiograph was performed for all patients for diagnosis and treatment planning purposes. Non-surgical periodontal treatment was done as needed. Impressions were taken and casted in stone for the fabrication of the surgical templates.

Surgical protocol As dictated by the randomization patients were assigned to either Buser's technique or to the VST. In the VST group, atraumatic tooth extraction was carried out using periotomes (Stoma, Storz am Mark GmbH, Emmingen-Liptingen Germany) under local anaesthesia (ARTINIBSA 4% 1:100.000. Inibsa Dental S.L.U. Barcelona, SPAIN).

Vestibular socket therapy (VST) included the following steps. a-traumatic tooth extraction, the socket curetted and rinsed with normal saline thoroughly. One-cm long vestibular access incision was made using a 15c blade (Stoma, Storz am Mark GmbH, Emmingen-Liptingen Germany) 3-4 mm apical to the mucogingival junction at the related socket . A subperiosteal tunnel was created connecting the socket orifice and the vestibular access incision using periotomes and micro periosteal elevators (Stoma, Storz am Mark GmbH, Emmingen-Liptingen Germany). Implant fixture (Biohorizons, Birmingham, Al, USA) were then inserted after drilling to its pre-planned location 3-4 mm apical to socket base with adequate primary stability achieved using a torque wrench reaching 30 Ncm torque . A flexible cortical membrane shield that is made of cortical bone of heterologous origin of 0.6 mm thickness (OsteoBiol® Lamina , Tecnoss®, Torino, Italy) was hydrated and then trimmed and introduced from the vestibular access incision reaching 1 mm below the socket orifice through the tunnel then stabilized using a membrane tack or a micro screw to the alveolar bone apical to the base of the socket (AutoTac System Kit, Biohorizons Implant Systems, Birmingham , Alabama Inc, USA) . The socket gap between the implant and the shield was then packed thoroughly with particulate bone graft (75% autogenous bone chips and 25% deproteinized bovine bone mineral (DBBM).

In Buser's group early implant placement, the failing tooth was extracted atraumatically using a periotome. A collagen plug was placed to stabilize the wound clot. A healing period of 4-8 weeks (depending on the size of the extracted tooth) was followed. Then an open flap implant surgery using a triangular flap design was cut. A slightly palatal incision in the edentulous area is done, with the incision made along the inner surface of the palatal bone wall deep into the socket allowing the entire regenerated soft tissue to be part of the buccal flap. After preparing the implant bed, the site was irrigated using normal saline. Implant was then placed under the crest of the palatal bone. A healing abutment was then attached.The bone graft was placed in a layered manner, where the cortical bone chips were placed first followed by the bio-oss activated mix. A non-cross liked membrane was then placed, after being soaked with BCM. Finally, the healing abutment was removed and the flap was released to allow for its suturing.

ELIGIBILITY:
Inclusion Criteria:

* all patients were adults ≥ 18 years
* 1-5 non-adjacent hopeless maxillary teeth in the esthetic zone.
* The involved teeth had type II sockets.
* To achieve optimum primary stability for the implants (30Ncm insertion torque), adequate palatal and at least 3 mm apical bone should be available to engage the immediately placed implants.

Exclusion Criteria:

* Smoking and/or pregnant patients
* systemic diseases
* a history of chemo- or radiotherapy within the past 2 years were excluded.
* Infected sockets were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
vertical and horizontal soft tissue changes | crown delivery and 1 year
  Amount of soft tissue changes were identified midfacially and at the apex of the mesial and distal papillae by superimposing the STL files of the models, obtained via intra-oral scanning, at the baseline (of the unrestorable tooth) with those after 12 months of implant insertion. The 3D software roughly aligned of both pre-and postoperative models through 3 identical points, identified on their surfaces. The best-fit algorithm of the software then perfected the superimposition process. The superimposed models were then imported into an STL viewer, where the measurements were performed. This method was proven to be accurate in volumetric measurements of hard and soft tissues.

SECONDARY OUTCOMES:
labial plate thickness changes | implant insertion -1 year
  Changes in the thickness of the labial plate of bone was measured by superimposing CBCT images obtained at the baseline (time of tooth extraction) and those after 12 months.
implant survival | Implant insertion- 1 year
  Implant survival was reported as defined by Buser et al by the absence of peri-implant infection, persistent subjective complaints such as pain, foreign body sensation, and/or dysesthesia, radiolucency around the implant, and/or any detectable implant mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Iman Radi, PhD, Study Director — Cairo University; AbdelSalam Alaskary, BDS, Principal Investigator — Private Practice
Locations (2):
- Egypt (2):
  - Faculty of dentistry, Cairo, Manial
  - ElAskary and Associates Private clinic, Alexandria

IPD SHARING:
Plan to Share IPD: No